CLINICAL TRIAL: NCT04849013
Title: Role of the Serotonin 5-HT2A Receptor in Mescaline-induced Altered States of Consciousness
Acronym: MDR
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: BASEC 2021-00035
Record Dates: First submitted 2021-03-26; First posted 2021-04-19 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Healthy
Keywords: Mescaline; Serotonin; Hallucinogen
MeSH Terms: interventions — Mescaline; Ketanserin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Placebo + Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Mescaline-100 + Placebo (Active Comparator)
  Interventions: Drug: Mescaline 100mg
- Mescaline-200 + Placebo (Active Comparator)
  Interventions: Drug: Mescaline 200mg
- Mescaline-400 + Placebo (Active Comparator)
  Interventions: Drug: Mescaline 400mg
- Mescaline-800 + Placebo (Active Comparator)
  Interventions: Drug: Mescaline 800mg
- Mescaline-800 + Ketanserin (Active Comparator)
  Interventions: Drug: Mescaline 800mg + Ketanserin 40mg

INTERVENTIONS:
Drug: Placebo — Drug: Placebo Capsules containing mannitol looking identical to the other drugs Other: Placebo Capsules containing mannitol looking identical to the other drugs
  Arms: Placebo + Placebo
Drug: Mescaline 100mg — Drug: 100mg Mescaline per os, single dose
  Other: Placebo (Capsules containing mannitol looking identical to the other drugs)
  Arms: Mescaline-100 + Placebo
Drug: Mescaline 200mg — Drug: 200mg Mescaline per os, single dose
  Other: Placebo (Capsules containing mannitol looking identical to the other drugs)
  Arms: Mescaline-200 + Placebo
Drug: Mescaline 400mg — Drug: 400mg Mescaline per os, single dose
  Other: Placebo (Capsules containing mannitol looking identical to the other drugs)
  Arms: Mescaline-400 + Placebo
Drug: Mescaline 800mg — Drug: 800mg Mescaline per os, single dose
  Other: Placebo (Capsules containing mannitol looking identical to the other drugs)
  Arms: Mescaline-800 + Placebo
Drug: Mescaline 800mg + Ketanserin 40mg — Drug: 800mg Mescaline per os, single dose
  Other: 40mg Ketanserin per os, single dose
  Arms: Mescaline-800 + Ketanserin

SUMMARY:
Mescaline (the active substance in Peyote and San Pedro cacti) is a classic and long known serotonergic psychedelic substance (hallucinogen) that is widely used for recreational, spiritual, and/or ethno medical purposes. Despite its long history, modern data on the acute effects of mescaline on human is lacking. Mescaline produces prototypical psychedelic effects, similar as lysergic acid diethylamide (LSD) and psilocybin. The serotonin 2A (5-HT2A) receptor is thought to primarily mediate acute alterations of consciousness induced by LSD and psilocybin. However, the contributory role of the 5-HT2A receptor in mescaline-induced alterations of consciousness is unclear. Using 5-HT2A receptor antagonist ketanserin, the psychedelic experience induced by LSD and psilocybin can be attenuated and shortened. The present study therefore explores the role the 5-HT2A receptor in mescaline-induced altered states of consciousness using escalating doses of mescaline and the 5-HT2A receptor blocker ketanserin administered before a high dose of mescaline.

Objective: The present MDR-study will characterize the subjective effects of different doses of mescaline using modern psychometric instruments and examine the contribution of the 5-HT2A receptor in the mescaline-induced alterations of consciousness.

Design: Double-blind, placebo-controlled, 6-period cross-over design with six treatment conditions. 1) Placebo (Pla + Pla), 2) 100 mg mescaline (Pla + 100mg mescaline), 3) 200 mg mescaline (Pla + 200mg mescaline), 4) 400 mg mescaline (Pla + 400mg mescaline), 5) 800 mg mescaline (Pla + 800mg mescaline), and 6) 40mg ketanserin and 800mg mescaline (Ket + 800mg mescaline).

Participants: 16 healthy participants aged ≥ 25 and ≤ 65 years (8 female, 8 male)

ELIGIBILITY:
Inclusion Criteria:

1. Age between 25 and 65 years old
2. Sufficient understanding of the German language
3. Understanding of procedures and risks associated with the study
4. Willing to adhere to the protocol and signing of the consent form
5. Willing to refrain from the consumption of illicit psychoactive substances during the study
6. Abstaining from xanthine-based liquids from the evenings prior to the study sessions to the end of the study days
7. Willing not to drive a traffic vehicle or operate heavy machinery within 48 hours after substance administration
8. Willing to use double-barrier birth control throughout study participation
9. Body mass index between 18-29 kg/m2

Exclusion Criteria:

1. Chronic or acute medical condition
2. Current or previous major psychiatric disorder
3. Psychotic disorder or bipolar disorder in first-degree relatives
4. Hypertension (>140/90 mmHg) or hypotension (SBP10 cigarettes/day)
5. Hallucinogenic substance use (not including cannabis) more than 20 times or any time within the previous two months
6. Pregnancy or current breastfeeding
7. Participation in another clinical trial (currently or within the last 30 days)
8. Use of medication that may interfere with the effects of the study medication
9. Tobacco smoking (>10 cigarettes/day)
10. Consumption of alcoholic beverages (>20 drinks/week)

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-08-11 (Actual); Primary Completion 2023-03-27 (Actual); Study Completion 2023-03-27 (Actual)

PRIMARY OUTCOMES:
Altered States of Consciousness | 18 months
  5 Dimensions of Altered States of Consciousness (5D-ASC) assesses mood, anxiety, derealization, depersonalization, changes in perception, auditory alterations, and reduced vigilance. The questionnaire is consisting of 94 items to be rated on a visual analog scale (horizontal line, 100 mm, marked with "not at all" on the left and "extremely" on the right), with higher values indicating stronger effects. Subjects will mark the scale with vertical lines.

SECONDARY OUTCOMES:
Extent of subjective response over time | 18 months
  Visual Analog Scales (VAS) will be repeatedly used to assess subjective alterations in consciousness over time. VAS will be presented as 100 mm long horizontal lines marked with "not at all" on the left and "extremely" on the right. The following VAS will be used: "any drug effect", "good drug effect", "bad drug effect", "stimulated", "happy", "anxiety", "nausea", "alteration of vision", "alterations of hearing", "sounds seem to influence what I see", "alteration of sense of time", "the boundaries between myself and my surroundings seem to blur", "I am having insights into connections that previously puzzled me", "open", "talkative", and "trust". Subjects will mark the scale with vertical lines.
Subjective mood ratings | 18 months
  Adjective Mood Rating Scale (AMRS) assesses the occurrence and intensity of 60 moods on a 4-point Likert scale ranging from "not at all" to "extremely".
Subjective experiences of spiritual phenomenons | 18 months
  Spiritual Realms Questionnaire (SRQ) assesses the spiritual phenomenons elicited by psychedelic substances through 11 main questions to be answered on a total of 65 sub-ordered visual analog scales (horizontal line, 100 mm, marked with "no, at all" on the left and "yes, very strong" on the right).
States of Consciousness | 18 months
  States of Consciousness Questionnaire (SCQ) assesses the emergence and intensity of phenomenons occurring in altered states of consciousness on a 6-point Likert scale ranging from 0 ("not at all") to 5 ("extremely").
Mystical-type experiences | 18 months
  Mystical-type experience questionnaire (MEQ) assesses with 30 items (embedded into the SCQ) the mystical experiences on a 6-point Likert scale ranging from 0 ("not at all") to 5 ("extremely").
Blood pressure | 18 months
  Blood pressure, assessed 20 times during each study session via systolic and diastolic blood pressure.
Heart rate | 18 months
  Heart rate, assessed 20 times during each study session via heart rate, Emax.
Body temperature | 18 months
  Body temperature assessed 20 times during each study session via tympanic body temperature.
Pupil size | 18 months
  Pupil size, assessed 8 times during each study session via pupilometer.
Mescaline concentrations in the blood | 18 months
  Mescaline and metabolites concentrations measured in the blood plasma, assessed 20 times during each study session via blood samples.
Mescaline concentrations in the urine | 18 months
  Mescaline and metabolites concentration measured in the urine, assessed in the total amount collected during each study session.
Effects on brain-derived neurotrophic factor (BDNF) | 18 months
  Plasma levels of brain-derived neurotrophic factor (BDNF), assessed 5 times during each study session via blood samples.
Effects on inflammatory cytokines | 18 months
  Plasma levels of INF-gamma, TNFalpha, Interleukins, assessed 5 times during each study session via blood samples.
Effects on oxytocin | 18 months
  Plasma levels of oxytocin, assessed 4 times during each study session via blood samples.
Emotional effects | 18 months
  Multifaceted Empathy Test (MET), effects on empathy in computer tests, assessed one time during each study session.
Effect moderation through personality traits I | 18 months
  Assessed one time during the screening via the NEO-Five-Factor-Inventory (NEO-FFI). The NEO-FFI assesses 5 personality traits (openness to experience, conscientiousness, extraversion, agreeableness and neuroticism) consisting of of 60 items. Each item is evaluated on a scale from -- "strong disagreement" to ++ "strong agreement".
Effect moderation through personality traits II | 18 months
  Assessed one time during the screening via Freiburger Personality Inventory (FPI). The FPI-R version comprises 138 items and covers 12 dimensions of personality: life satisfaction, social orientation, performance orientation, inhibition, excitability, aggressiveness, stress, physical complaints, health concerns, openness, as well as the secondary factors according to Eysenck's Extraversion and Emotionality (Neuroticism). It uses a 2-point scale ("true" and "not true").
Effect moderation through personality traits III | 18 months
  Assessed one time during the screening via Saarbrücker Personality Questionnaire (SPF). The SPF defines empathy as the "reactions of one individual to the observed experiences of another." It assesses 28-items on a 5-point Likert scale ranging from "Does not describe me well" to "Describes me very well". The measure has 4 subscales (Perspective Taking, Fantasy, Empathic Concern, Personal Distress) each made up of 7 different items.
Effect moderation through personality traits IV | 18 months
  Assessed one time during the screening via HEXACO personality inventory (Honesty-Humility, Emotionality, Extraversion, Agreeableness, Conscientiousness, and Openness). The HEXACO consists of 100 items. Each item is evaluated on a scale from 1 "strong disagreement" to 5 "strong agreement".
Effect moderation through personality traits V | 18 months
  Assessed one time during the screening via Defense Style Questionnaire (DSQ-40). The DSQ-40 can provide scores for 20 individual defenses, and scores for the three factors "mature", "neurotic", and "immature". Each item is evaluated on a scale from 1 to 9, where "1" indicates "completely disagree" and "9" indicates "fully agree".
Psychological insight | 18 months
  Psychological insight questionnaire (PIQ), assesses painful insights during a psychedelic experience with 14 items (6-point Likert scale ranging from 0 ("not at all") to 5 ("extreme/more than ever before")).
Effects on life satisfaction, well-being and appreciation I | 18 months
  Scale of Positive and Negative Experience (SPANE), assesses life satisfaction regarding the preceding week with12 items (5-point Likert scale ranging from 1 ("very rarely") to 5 ("very often")).
Effects on life satisfaction, well-being and appreciation II | 18 months
  Berner Subjective Well-Being Questionnaire for Adolescents (BFW/E), assesses optimism with 8 items (6-point Likert scale ranging from 1 ("completely wrong") to 6 ("completely right")).
Effects on life satisfaction, well-being and appreciation III | 18 months
  Global Life Satisfaction (GLS), assesses life satisfaction with a single question (ranging from 0 ("not at all satisfied") to 10 ("entirely satisfied")).
Effects on life satisfaction, well-being and appreciation IV | 18 months
  Appreciation Scale (AS), assesses appreciation with 57 questions (7-point Likert scale ranging from 1 ("never") to 7 ("several times a day")).
Incidence of Adverse Events before and during each study session | 18 months
  Major adverse events concerning the subject's health during study inclusion (if present) are registered by semi-structured interviews.
Incidence of Adverse Events during each study session | 18 months
  List of complaints (LC), which covers the emergence of 66 complaints in a yes/no format, assessed three times during each study session.
Electrical activity of the heart | 18 months
  Electrocardiogram (ECG) will be recorded twice during the study sessions (baseline and at peak drug effect) as well as on the screening exam to assess potential drug effects on the QTc interval.

CONTACTS AND LOCATIONS:
Overall Officials: Matthias E Liechti, Prof. Dr. MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Clinical Trial Unit, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mueller L, Klaiber A, Ley L, Becker AM, Thomann J, Luethi D, Schmid Y, Liechti ME. Pharmacokinetics, Pharmacodynamics, and Urinary Recovery of Oral Mescaline Hydrochloride in Healthy Participants. Clin Pharmacokinet. 2025 Oct;64(10):1495-1506. doi: 10.1007/s40262-025-01544-x. Epub 2025 Jul 14. PMID 40658345